CLINICAL TRIAL: NCT00518583
Title: A Phase II Study of Pre-Operative Pegylated Liposomal Doxorubicin (PLD), Paclitaxel, and Trastuzumab in Patients With Operable Breast Cancer Over-expressing Her2-neu
Brief Title: Phase II Study in Patients With Operable Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aptium Oncology Research Network (Network)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Responsible Party: Marti McKinley, Aptium Oncology Research Network
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06BR01
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Over-expressing Her2-neu
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin (Doxil) — Doxorubicin administered once every three weeks Taxol administered weekly Herceptin administered weekly
  Other Names: taxol (paclitaxel); herceptin

SUMMARY:
The study will evaluate the safety and efficacy of the combination PLD, paclitaxel, and trastuzumab in patients with operable breast cancer. Patients will be treated with the combination for 18 weeks, followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Dx of clinical T1c-T3, N0-1, M0 breast cancer
* Interval between diagnosis and consent of <- 62 days
* Life expectancy of 10 years
* LVEF by MUGA >= lower limit of normal for the testing facility
* Negative serum pregnancy test
* Adequate bone marrow, renal, liver function
* Negative bone scan
* HRT discontinued before study entry
* Adequate contraceptive methods

Exclusion Criteria:

* Male breast cancer
* Less than 21 years of age
* Ulceration, infiltration of the skin, complete fixation or severe skin edema
* N3 disease in which nodes are matted and fixed
* Suspicious palpable supraclavicular nodes
* CT evidence of malignant internal mammary nodes
* Pregnancy or breast feeding at time of study entry
* Prior therapy for breast cancer
* Prior anthracycline for any malignancy
* Prior breast malignancy of the contralateral breast
* Prior non-breast malignancy within 5 years
* Non-malignant disease that would preclude follow up
* MI within 6 months, NYHA Class II or greater heart failure
* Psychiatric disorders or conditions that would preclude provision of informed consent

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-01 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Identify the pCR rate of neoadjuvant chemotherapy using the proposed 18-week regimen of PLD + paclitaxel + trastuzumab | within 18 weeks

SECONDARY OUTCOMES:
Identify the complete response rate | within 18 weeks
Identify the partial response rate | within 18 weeks
Identify the overall response rate | within 18 weeks
Evaluate changes in cardiac function | within study participation
Monitor safety and tolerability of neoadjuvant chemotherapy using the proposed 18 week regimen | within study participation

CONTACTS AND LOCATIONS:
Overall Officials: John Macdonald, MD, Study Director — CMO Aptium Oncology
Locations (9):
- United States (9):
  - Providence St. Joseph Medical Hospital, Burbank, California
  - Cedars-Sinai Outpatient Cancer Center, Los Angeles, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Lynn Regional Cancer Center West, Boca Raton, Florida
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Maimonides Cancer Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - St Vincent Comprehensive Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio